CLINICAL TRIAL: NCT06676371
Title: Randomized Control Trial of Total Arch Replacement With Frozen Elephant Trunk Versus Conventional Hemiarch Replacement in Patients With Acute Type A Aortic Dissection (TARFET-TAAD)
Brief Title: Total Arch Replacement With Frozen Elephant Trunk Versus Hemiarch Replacement in the Management of Acute Type A Aortic Dissection
Acronym: TARFET-TAAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: University of Vienna (Other); Mahidol University (Other)
Responsible Party: Principal Investigator, Randolph Wong, Professor and Chief of Division of Cardiothoracic Surgery, Department of Surgery, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRER Ref No.: NTEC-2024-574
Record Dates: First submitted 2024-10-28; First posted 2024-11-06 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-10

CONDITIONS: Aortic Dissection Type A
Keywords: Total Arch Replacement and Frozen Elephant Trunk (TARFET); Conventional Hemiarch (HAR) replacement; Acute Type A aortic dissection (ATAAD)

STUDY DESIGN:
Intervention Model Description: Randomized control trial of two groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Hemiarch group (HAR) (Active Comparator): Under general anesthesia and transesophageal echocardiogram monitoring, a median sternotomy will be performed. Patients will be placed on cardiopulmonary bypass using arterial inflow from the femoral artery, axillary artery, or direct aortic cannulation, along with right atrial appendage venous cannulation. Systemic cooling to 25 degrees Celsius will commence, followed by thiopental coma and circulatory arrest. The aorta will be trimmed to the distal ascending aorta or proximal arch, and antegrade cerebral perfusion will be initiated to the brachiocephalic branch.
  The distal anastomosis will connect a vascular graft to the distal ascending aorta or aortic arch. After completing this, systemic perfusion and rewarming will begin, followed by the proximal anastomosis with the vascular graft. After de-airing, the aorta will be de-clamped, and the patient will be weaned from cardiopulmonary bypass and decannulated. Hemostasis and sternal closure will follow standard institutional protocols
  Interventions: Procedure: Conventional hemiarch replacement
- Total Arch Replacement and Frozen Elephant Trunk group (TARFET) (Active Comparator): Under general anesthesia and transesophageal echocardiogram monitoring, a median sternotomy will be performed. Patients will be placed on cardiopulmonary bypass via femoral, axillary, or direct aortic cannulation. Systemic cooling to 25 degrees Celsius will lead to thiopental coma and circulatory arrest. The aorta will be trimmed to the distal arch, with antegrade cerebral perfusion initiated.
  Distal anastomosis will connect a vascular graft to the distal arch, followed by visceral perfusion, rewarming, and proximal anastomosis. After de-airing, the aorta will be de-clamped, and the patient will be weaned from bypass and decannulated. Hemostasis and sternal closure will follow standard protocols.
  Arterial cannulation sites for HAR and TARFET will be determined by the surgeon based on the clinical scenario.
  Interventions: Procedure: E-vita® Open Neo; Artivion; Procedure: Thoraflex Hybrid; Terumo

INTERVENTIONS:
Procedure: Conventional hemiarch replacement — Conventional open hemiarch replacement
  Arms: Conventional Hemiarch group (HAR)
Procedure: E-vita® Open Neo; Artivion — E-vita® Open Neo is a hybrid stent graft system for aortic arch and descending thoracic aorta repair with Frozen Elephant Trunk Technique.
  Arms: Total Arch Replacement and Frozen Elephant Trunk group (TARFET)
Procedure: Thoraflex Hybrid; Terumo — The Thoraflex Hybrid is a device system designed to repair a weakened and bulging section (aneurysm) and/or a tear in the lining (dissection) of the aorta behind the heart (aortic arch). The system includes a polyester graft section that reinforces a weakened section of the blood vessel, a connected stented section (nitinol wire frame on polyester graft material) that holds the artery open, and a delivery catheter that is used to place the device. The polyester graft and stented sections are coated with a protein substance taken from animal body parts (gelatin) to seal the implant and prevent blood from leaking out.
  Arms: Total Arch Replacement and Frozen Elephant Trunk group (TARFET)

SUMMARY:
Acute Type A aortic dissection (ATAAD) and its complications are life-threatening conditions that cause more than 1400 hospital admissions and 300 deaths every year in Hong Kong and cause 172,927 deaths globally in 2019. There is an increasing trend in recent years.

Given the hyperacute presentation and complexity of the clinical manifestation with various mal-perfusion syndromes, the mortality of ATAAD remained high in all international reported registries and published series.

Conventional Hemiarch (HAR) replacement has been the gold standard procedure for ATAAD in most of cardiac surgical centers around the world because of the relative simplicity of the procedure. However, around 50-70% of patients were reported to develop distal anastomosis new entry after hemiarch procedure and for those with entry tear over aortic arch and distal mal-perfusion, hemiarch alone might not be able to solve the downstream problem. On the other hand, total arch replacement and frozen elephant trunk procedure (TARFET) is more complex, technically demanding procedure that could potentially cover/resect the arch entry tear and exclude tear over proximal descending thoracic aorta and, hence, solve the distal mal-perfusion syndrome. To date, there is no randomized control trial to answer whether HAR or TARFET procedure is superior in patients with ATAAD and entry tear is over the aortic arch or proximal descending thoracic aorta.

We plan to conduct a multi-center trial to recruit consecutive patients with ATAAD with entry tear beyond ascending aorta and randomized them, after informed consent, into either the conventional hemiarch replacement group (HAR) or total arch replacement and frozen elephant trunk (TARFET). The participating centers will collect pre- operative, intra-operative and post-operative clinical parameters for two groups of patients via REDCap system. Written informed consent, specifically allowing the use of clinical records for this randomized study, will be obtained from every patient prior to data collection. The primary outcome is the 30-day mortality of the ATAAD patients with surgically treated by HAR versus TARFET approach. The secondary outcomes are the major adverse cardiovascular and cerebral events, post-op renal replacement therapy, re-exploration for bleeding and re-intervention within 30-days.

This study will be the world's first multi-center randomized control trial in ATAAD to compare the 30-day mortality of patients treated with HAR and TARFET. It could be a guideline-changing study for the treatment of ATAAD and its impact on the surgical approach to patients suffering from ATAAD.

DETAILED DESCRIPTION:
Project Objectives:

1. The primary objective is to evaluate the all-cause 30-day mortality rate between the TARFET and HAR groups in patients with acute type A aortic dissection with entry tear beyond ascending aorta.
2. The secondary objective is to evaluate the impact of TARFET and HAR in patients with ATAAD complicated with mal-perfusion syndrome.
3. The third objectives include comparing the rates of major adverse cardiovascular and cerebrovascular events (MACCE), renal replacement therapy, aortic reintervention, and other relevant clinical outcomes within 30 days.

Background Acute Type A aortic dissection (ATAAD) and its complications are life-threatening conditions that cause more than 1400 hospital admissions and 300 deaths every year in Hong Kong and cause 172,927 deaths globally in 2019. There is an increasing trend in recent years. Given the hyperacute presentation and complexity of the clinical manifestation with various mal-perfusion syndromes, the mortality of ATAAD remained high in all international reported registries and published series. (IRAD and GERAAD). For the same reason, high quality clinical studies are lacking, and the current guideline are largely based on non-randomized clinical trials and prospective studies (EACTS/STS/AHA guideline). Data from international registries showed the mortality of surgically treated ATAAD was around 17-26% and those with mal-perfusion had even higher mortality. The primary goals of surgical therapy in ATAAD are to replace the ascending thoracic aorta together with the primary entry tear, sealing of the false lumen (FL) and the distal anastomotic site and decompression the false lumen and resolve distal mal-perfusion. Conventional Hemiarch (HAR) replacement has been the gold standard procedure for ATAAD in most of cardiac surgical centers around the world because of the relative simplicity of the procedure. However, around 50-70% of patients were reported to develop distal anastomosis new entry (DANE) after hemiarch procedure and for those with entry tear over aortic arch and distal mal-perfusion, hemiarch alone might not be able to solve the downstream problem. On the other hand, total arch replacement and frozen elephant trunk procedure (TARFET) is a more complex and technically demanding procedure that could potentially cover/resect the arch entry tear and exclude tear over proximal descending thoracic aorta and, hence, solve the distal mal-perfusion syndrome. To date, there is no randomized control trial to answer whether HAR or TARFET procedure is superior in patients with ATAAD where entry tear is beyond ascending aorta. The investigators aim to conduct a multi-centers, randomized control trial to compare the 30-day mortality of patients with ATAAD who undergo HAR versus TARFET.

Main research questions

1. To evaluate the all-cause 30-day mortality rate between the TARFET and HAR groups in patients with ATAAD where entry tear is beyond the ascending aorta.
2. To evaluate the impact of TARFET and HAR in patients with ATAAD complicated with mal-perfusion syndrome.
3. To compare the rates of major adverse cardiovascular and cerebrovascular events (MACCE), renal replacement therapy, aortic reintervention, and other relevant clinical outcomes.

Hypothesis In ATAAD with entry tear beyond ascending aorta with or without mal-perfusion, there is no survival benefit by performing TARFET when compared with HAR

Study Design:

This will be a multi-center, randomized controlled trial to compare the clinical outcomes of HAR and TARFET in patients with acute aortic dissection with entry tear(s) beyond ascending aorta.

Centers involved

1. Division of Cardiothoracic Surgery, Department of Surgery, Prince of Wales Hospital, the Chinese University of Hong Kong, Hong Kong SAR
2. Department of Cardiac Surgery, Faculty of Medicine, University of Vienna, Austria: Co- I: Prof Marek Erhlich
3. Division of Cardiothoracic Surgery, Siriraj Hospital, Faculty of Medicine, Mahidol University, Thailand: Co-I: Prof Worawong Slisatkorn

Inclusion and Exclusion criteria:

Consecutive patients with acute thoracic aortic dissection diagnosed within 2 weeks of the onset of the symptoms with the diagnosis made by CT scan will be screened.

Methodology:

In this study, the investigators plan to prospectively recruit consecutive patients with ATAAD with entry tear beyond ascending aorta and randomized them, after informed consent, into either the HAR or TARFET group. The participating team will collect pre-operative, intra-operative, and post- operative clinical and radiological parameters for two groups of patients. Written informed consent, specifically allowing the use of clinical records for this randomized study, will be obtained from every patient prior to data collection. Patient data will be documented at the following time points: Pre-operative, intervention(s), discharge(s) from the hospital. Source data verification will be performed on 100% of the patients; data in the database will be reviewed and verified against existing source documents by a dedicated research assistant. Complete DICOM image files of the CT scans will be evaluated by site Investigator to ascertain the patients fulfilled the radiological inclusion criteria.

Study population Screening and randomization A computer-generated randomization sequence will be generated by the research assistant using the online randomization software. A total of 150 patients will be randomized 1:1 to one of the two treatment arms. Block randomization with block size of 8 is used to maintain good balance to each treatment group. The randomization list will be kept in a set of tamper-evident envelopes. The envelopes will be identical and sealed. The trial identifier with a sequential number will be printed on each envelope and the inside will contain the treatment allocation. Envelopes will be unsealed by the on-call surgeon to reveal the allocation treatment prior to the surgery.

Patients, with their consent, will be recruited to participate by investigators after considering the inclusion and exclusion criteria.

Blinding of the study After randomization, the recruited patient will be allocated to either HAR or TARFET group. There will be no blinding of the randomization result to the recruited patients, the operating surgeons, and the clinician-in-charge.

Treatment Procedures

Conventional Hemiarch group (HAR):

Under general anesthesia and trans-esophageal echocardiogram monitoring, a median sternotomy will be performed. Patients will be put on cardiopulmonary bypass with arterial inflow from femoral artery/axillary artery/direct aortic cannulation and right atrial appendage venous two-stage cannulation. Systemic cooling to 25 Degree Celsius will commence. At a temperature of 25 Degree Celsius and thiopentone coma, the circulatory arrest will begin. The aorta will be trimmed to the level of the distal ascending or proximal arch. Antegrade cerebral perfusion will be started to the brachiocephalic branch of the aortic arch. The distal anastomosis will be done between a vascular graft and the distal ascending aorta/aortic arch. After the distal anastomosis is completed, visceral and cerebral systemic perfusion and rewarming will be started. The proximal ascending aorta will be anastomosed with the proximal end of the vascular graft. After de-airing and aorta will be de-clamped and the patient will be weaned from cardiopulmonary bypass and decannulated. Hemostasis and sternal closure will be done as per routine protocol of the individual institution.

Total Arch Replacement and Frozen Elephant Trunk group (TARFET):

Under general anesthesia and trans-esophageal echocardiogram monitoring, a median sternotomy will be performed. Patients will be put on cardiopulmonary bypass with arterial inflow from femoral artery/axillary artery/direct aortic cannulation and right atrial appendage venous two-stage cannulation. Systemic cooling to 25 Degree Celsius will commence. At a temperature of 25 Degree Celsius and thiopentone coma, the circulatory arrest will begin. The aorta will be trimmed to the level of the distal arch. Antegrade cerebral perfusion will be started to the brachiocephalic, left common carotid and left subclavian branches of the aortic arch. The distal anastomosis will be done between a vascular graft and the distal arch at zone 2 or zone 3 at the discretion of the operating surgeon. After the distal anastomosis is completed, visceral systemic perfusion and rewarming will be started. The proximal ascending aorta will be anastomosed with the proximal end of the vascular graft followed by individual head and neck vessels perfusion. After de-airing and aorta will be de-clamped and the patient will be weaned from cardiopulmonary bypass and decannulated. Hemostasis and sternal closure will be done as per routine protocol of the individual institution.

The exact arterial cannulation site(s) for HAR and TARFET will be at the discretion of the operating surgeon according to the clinical scenario and intra-operative findings. These parameters will be recorded and analysed accordingly.

Perioperative management The perioperative management of all recruited patients is standardized. All patients receive prophylactic antibiotics during induction and until all drains are removed in the postoperative period. All patients will have invasive blood pressure monitoring with an arterial line and intravenous antihypertensive medications aiming to control systolic blood pressure to below 140mmHg.

Randomization:

Eligible patients will be randomized 1:1 to the TARFET or HAR group using a computerized, permuted-block randomization scheme, stratified by site. The randomization sequence will be generated by an independent statistician and concealed from the study team. Screening log will also be kept by the individual institution.

Data Management and Analysis:

All data will be collected and managed using a secure, web-based electronic data capture system.

An independent Data and Safety Monitoring Board (DSMB) will regularly review the study data and safety outcomes and make recommendations to the Steering Committee.

The primary analysis will be conducted on an intention-to-treat basis, comparing the 30-day all-cause mortality rates between the two groups using a Chi-square test. Secondary analyses will evaluate the other clinical outcomes.

Ethical consideration:

This study shall be conducted in accordance with the ethical principles in the Declaration of Helsinki. This protocol will be submitted to the Clinical Ethical Review Committees (CREC) of individual institution for approval. The clinical investigation shall not begin until CREC approval has been obtained. Any additional requirements imposed by the CREC shall be followed. Written informed consent, specifically allowing the use of clinical records for study purposes, will be obtained from every patient prior to data collection. Patients can withdraw from the study without any prejudice at any time during the study. Data will be kept confidential in secure offices/location of the Department of Surgery of corresponding institution for seven years.

Confidentiality:

All laboratory specimens, evaluation forms, reports, and other records will be stored de- identified with a unique study ID to maintain research participant confidentiality. All clinical records will be kept in a secure storage area in the Department of Surgery of the corresponding institutions. Clinical information will not be released without the written permission of the research participant except as necessary for monitoring by regulatory bodies, and/or the IRB/EC.

The Investigators and all employees and research staff involved with this study may not disclose or use any data, record, or other unpublished, confidential information for any purpose other than performance of the study.

Potential risks of the study:

Acute aortic dissection is a life-threatening emergency condition with mortality of around 18- 25% from the world registries. In both the P-I and Co-I units, the investigators can achieve 30-days mortality of less than 20% from the previously published series. The study team should carefully assess the risks associated with each surgical intervention and implement strategies to minimize these risks, such as stringent patient selection criteria, meticulous surgical techniques, and robust perioperative management protocols. The potential benefits of the study interventions, including improved survival and reduced complications, should be clearly communicated to the participants. The study design should aim to maximize the potential benefits to the participants and future patients, while minimizing the risks. The investigators believe there will be minimal risk incur to the study patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient 's age is between 18 and 80 years.
2. Patient is willing and able to give informed consent.
3. Patient has acute type A aortic dissection with entry tear beyond ascending aorta.
4. Patient not in coma/irreversible end organ failure/cardiac massage for resuscitation

Exclusion Criteria:

1. There is no identifiable entry tear in the aorta
2. The ascending entry tear extends into aortic arch
3. Patient has entry tear only in ascending aorta
4. Patient with Type B aortic dissection
5. Patient has co-morbidity (i.e. active malignancy (progressive, stable or partial remission)) causing expected survival to be less than 2 years.
6. Patient has any other medical, social, or psychological problems, that in the opinion of the investigator, preclude the patient from participating in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the all-cause 30-day mortality rate between the TARFET and HAR groups in patients with acute type A aortic dissection with entry tear beyond ascending aorta. | From enrollment to the end of treatment at 30 days

SECONDARY OUTCOMES:
Malperfusion with respect to radiological evidence | From enrollment to 12 months after treatment.
  True lumen cross sectional area divided by total aortic cross sectional area at the narrowest part in descending thoracic aorta.
  Significant radiological ischemia definited as <20% (True Lumen/Total aortic cross sectional area)
Malperfusion with respect to biochemical evidence | From enrollment to 12 months after treatment.
  High lactate: Lactate > 4
Malperfusion with respect to biochemical evidence | From enrollment to 12 months after treatment.
  Acidosis: pH < 7.35
Malperfusion with respect to biochemical evidence | From enrollment to 12 months after treatment.
  Dearranged LFT: any increase in ALP, ALT, Bilirubin 5% more than baseline
Malperfusion with respect to biochemical evidence | From enrollment to 12 months after treatment.
  Derranged RFT: any increase in Cr 5% more than baseline
Malperfusion with respect to biochemical evidence | From enrollment to 12 months after treatment.
  Increased LDH: increase more than normal range
Malperfusion with respect to biochemical evidence | From enrollment to 12 months after treatment.
  Increased myoglobin: increase more than normal range
Malperfusion with respect to clinical evidence | From enrollment to 12 months after treatment.
  Absent or weakness of pulse
Malperfusion with respect to clinical evidence | From enrollment to 12 months after treatment.
  Limb weakness (modified Rankin Scale (mRS)) No symptoms (0), no significant disability; able to carry out all usual activities, despite some symptoms (1), slight disability; able to look after own affairs without assistance, but unable to carry out all previous activities (2), moderate disability; requires some help, but able to walk unassisted (3), moderately severe disability; unable to attend to own bodily needs without assistance, and unable to walk unassisted (4), Severe disability; requires constant nursing care and attention, bedridden, incontinent (5) left, right, both / time point of last event
Malperfusion with respect to clinical evidence | From enrollment to 12 months after treatment.
  Paraplegia or paraparesis (modified Tarlov score) No lower extremity movement (0, paraplegia), lower extremity motion without gravity (1, paraplegia), Lower extremity motion against gravity (2, paraplegia), able to stand with assistance (3 paraparesis), able to walk with assistance (4, paraparesis), normal (5, normal)

OTHER OUTCOMES:
Percentage of patients with Major Adverse Events | From enrollment to the end of treatment at 30 days
  Rate of patients who are free from the following Major Adverse Events (MAEs) (new permanent disabling stroke), new permanent (> 30 days) paraplegia or paraparesis, reintervention (excluding reoperation for bleeding or planned or unplanned additional intervention), visceral mal-perfusion, limb(s) ischemia
Percentage of patients requiring additional aortic intervention | From enrollment to the end of treatment at 30 days
  Rate of patients with aortic rupture and additional intervention (planned / unplanned)
Percentage of patients with Renal failure | From enrollment to the end of treatment at 30 days
  Renal failure requiring permanent (> 90 days) dialysis or hemofiltration in a patient with a normal pre-procedure serum creatinine level

CONTACTS AND LOCATIONS:
Locations (3):
- University Hospital Vienna, Vienna, Austria
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Siriraj Hospital - Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Anonymized clinical and radiological outcome data will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available when we complete our analysis and for a 12-month period
Access Criteria: Approval needs to be sought from the Principal Investigator

REFERENCES:
- [Background] Lombardi JV, Hughes GC, Appoo JJ, Bavaria JE, Beck AW, Cambria RP, Charlton-Ouw K, Eslami MH, Kim KM, Leshnower BG, Maldonado T, Reece TB, Wang GJ. Society for Vascular Surgery (SVS) and Society of Thoracic Surgeons (STS) Reporting Standards for Type B Aortic Dissections. Ann Thorac Surg. 2020 Mar;109(3):959-981. doi: 10.1016/j.athoracsur.2019.10.005. Epub 2020 Jan 27. PMID 32000979
- [Background] Ho JYK, Kim CH, Chow SCY, Kwok MWT, Lee H, Kim TH, Fujikawa T, Wong RHL, Song SW. Initial Asian experience of the branched E-vita open NEO in complex aortic pathologies. J Thorac Dis. 2023 Feb 28;15(2):484-493. doi: 10.21037/jtd-22-1055. Epub 2023 Feb 22. PMID 36910067
- [Background] Fujikawa T, Kwok M, Ho J, Wong R. Open descending aortic replacement after Thoraflex hybrid graft implantation. Multimed Man Cardiothorac Surg. 2020 Jan 27;2020. doi: 10.1510/mmcts.2020.004. PMID 32191402
- [Background] Tsagakis K, Kempfert J, Zierer A, Martens A, Dohle DS, Castiglioni A, Wong RH, Widenka K, Liakopoulos O, Borger MA, Oo AY, Holubec T, Luehr M, Legarra Calderon JJ, Grabenwoger M. E-vita OPEN NEO in the treatment of acute or chronic aortic pathologies: first interim results of the NEOS study. Eur J Cardiothorac Surg. 2024 Jun 3;65(6):ezae206. doi: 10.1093/ejcts/ezae206. PMID 38830042
- [Background] Rylski B, Hahn N, Beyersdorf F, Kondov S, Wolkewitz M, Blanke P, Plonek T, Czerny M, Siepe M. Fate of the dissected aortic arch after ascending replacement in type A aortic dissectiondagger. Eur J Cardiothorac Surg. 2017 Jun 1;51(6):1127-1134. doi: 10.1093/ejcts/ezx062. PMID 28369453
- [Background] Czerny M, Schoenhoff F, Etz C, Englberger L, Khaladj N, Zierer A, Weigang E, Hoffmann I, Blettner M, Carrel TP. The Impact of Pre-Operative Malperfusion on Outcome in Acute Type A Aortic Dissection: Results From the GERAADA Registry. J Am Coll Cardiol. 2015 Jun 23;65(24):2628-2635. doi: 10.1016/j.jacc.2015.04.030. PMID 26088302
- [Background] Hagan PG, Nienaber CA, Isselbacher EM, Bruckman D, Karavite DJ, Russman PL, Evangelista A, Fattori R, Suzuki T, Oh JK, Moore AG, Malouf JF, Pape LA, Gaca C, Sechtem U, Lenferink S, Deutsch HJ, Diedrichs H, Marcos y Robles J, Llovet A, Gilon D, Das SK, Armstrong WF, Deeb GM, Eagle KA. The International Registry of Acute Aortic Dissection (IRAD): new insights into an old disease. JAMA. 2000 Feb 16;283(7):897-903. doi: 10.1001/jama.283.7.897. PMID 10685714
- [Background] Hospital Authority Statistical Report 2011-2012, Page 30, Table 1.2 www.ha.org.hk/upload/publication_15/471.pdf
- [Background] Hospital Authority Statistical Report 2009-2010, Page 28, Table 1.1 www.ha.org.hk/upload/publication_15/321.pdf
- [Background] Centre for Health Protection, Vital Statistics, Death Rates by Leading Causes of Death 1981-2000 www.chp.gov.hk/en/data/4/10/27/115.html
- See also: Sample size calculator — https://clincalc.com/stats/SampleSize.aspx
- See also: Total Aortic Arch Replacement — https://www.youtube.com/watch?v=BcwykNGsTlU